CLINICAL TRIAL: NCT00311805
Title: Injection of Autologous CD34-Positive Stem Cells for Neovascularization and Symptom Relief in Patients With Severe Intermittent Claudication
Brief Title: Autologous CD34+ Stem Cell Injection for Severe Intermittent Claudication (Leg Pain)
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Losordo, Douglas, M.D. (Individual)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STU00023438/STU00000487; 11931-01 (Other: Sponsor protocol number)
Record Dates: First submitted 2006-04-04; First posted 2006-04-06 (Estimated); Last update posted 2015-03-31 (Estimated); Status verified 2015-03

CONDITIONS: Peripheral Artery Disease; Severe Intermittent Claudication
MeSH Terms: conditions — Peripheral Arterial Disease; Intermittent Claudication | interventions — Antigens, CD34

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator)
  Interventions: Biological: Autologous Stem Cells (CD34+)
- 2 (Active Comparator)
  Interventions: Biological: Autologous Stem Cells (CD34+)
- 3 (Placebo Comparator)
  Interventions: Biological: Autologous Stem Cells (CD34+)

INTERVENTIONS:
Biological: Autologous Stem Cells (CD34+) — Intramuscular Injections

SUMMARY:
The goal of the study is to determine the safety and possible effectiveness of various doses of autologous (one's own) stem cells, delivered with a needle into the regions of the leg with poor blood flow in patients with blocked leg arteries that results in claudication (pain when walking). Stem cells are primitive cells produced by the bone marrow that can develop into blood cells or other types of cells. In addition to determining whether this new approach is safe, the diagnostic tests may offer preliminary insights into the usefulness of this approach for treating intermittent claudication - the condition where areas in the leg are lacking enough oxygen and blood flow to keep the leg muscle working well, causing pain and cramping upon walking.

This study is a double-blind, randomized study to compare CD34-positive stem cells versus a placebo agent (salt water solution known as normal saline). The patient will have a 3:1 chance of their stem cells versus the placebo. Regardless of a patient receiving placebo or treatment, all patients will undergo all of the pre-treatment phases of this study, which includes the stem cell mobilization and apheresis procedure.

ELIGIBILITY:
Inclusion Criteria:

* Males or females equal to or greater than 21 years old
* Patients with infra-inguinal atherosclerosis with a stenosis or occlusion of a major vessel in the affected limb(s) of one or more of the following arteries: superficial femoral, popliteal, or one or more infrapopliteal arteries, which is/are non-reconstructable.
* Patients with symptoms of Severe Intermittent Claudication in at least 1 lower limb persisting for at least 6 months (Rutherford Class 3).
* Patients who have a diagnosis of Peripheral Arterial Disease (PAD) in at least 1 lower limb secondary to atherosclerosis, for at least 6 months.

Exclusion Criteria:

* Patients who have had successful aortic or lower extremity arterial surgery, angioplasty, or lumbar sympathectomy within 3 month preceding screening.
* Patients with iliac disease amenable to revascularization.
* Patients judged to be a suitable candidate for surgical or percutaneous revascularization in the limb in which treatment is proposed.
* Patients with Critical Limb Ischemia (CLI), Rutherford Symptom Score of 4,5, or 6.
* Patients in who arterial insufficiency in the lower extremity is the result of a non-atherosclerotic disorder.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2006-04; Primary Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Safety of Intramuscular administration of CD34-positive cells | All

SECONDARY OUTCOMES:
Functional improvement | Week 12, Month 6, Month 12

CONTACTS AND LOCATIONS:
Overall Officials: Douglas W. Losordo, M.D., Principal Investigator — Northwestern University
Locations (2):
- United States (2):
  - Cardiology, PC, Birmingham, Alabama
  - Northwestern University, Chicago, Illinois